CLINICAL TRIAL: NCT01111500
Title: First Time Anterior Glenohumeral Joint Dislocation With a Bankart Lesion in Young Patients: Which Type of Immobilization Should be Chosen? A Prospective Randomized Study
Brief Title: Immobilization After an Anterior Glenohumeral Joint Dislocation With a Bankart Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEJ-399
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Glenohumeral Joint Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- external rotation immobilization (Active Comparator): Patient will wear an external rotation brace to immobilize the injured arm.
  Interventions: Device: Donjoy ER brace
- internal rotation immobilization (Active Comparator): Patient will wear an internal rotation brace to immobilize the injured arm.
  Interventions: Device: Thoraco brachial brace

INTERVENTIONS:
Device: Donjoy ER brace — Patients will wear an external rotation brace, the Donjoy ER brace, during treatment.
  Arms: external rotation immobilization
Device: Thoraco brachial brace — Patients will wear an internal rotation brace, a thoraco brachial brace, during treatment.
  Arms: internal rotation immobilization

SUMMARY:
Glenohumeral joint dislocation is the most frequent joint dislocation with a prevalence of 1.7/100000 citizens/year. It is treated by reduction, under sedation or anaesthesia, followed by an immobilization of the arm.

The purpose of the study is to evaluate the healing of the labrum in first time anterior glenohumeral joint dislocation with a Bankart lesion in young patients by comparing an external rotation brace to an internal rotation brace to immobilize the injured arm.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* < 40 years old
* anterior glenohumeral joint dislocation proved by radiography
* dislocation needing a reduction manoeuvre
* home close to evaluation site for 24 months follow-up visits
* signed consent form

Exclusion Criteria:

* associated fracture
* Hill-Sachs lesion = or > than 30%
* neurovascular deficit
* hypermobility
* pre-existing instability of the injured shoulder
* systemic neurological disease
* allergy to gadolinium
* functional sequel to the shoulder due to previous injury
* incapacitated adult patient
* minor patient
* home far from evaluation site
* refusal to sign the consent form

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-07; Primary Completion 2013-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Anatomical healing of the labrum | 3 months after dislocation
  An MRI with usual cuts in ABER and ADIR positions are performed to demonstrate the anatomical healing of the labrum.

SECONDARY OUTCOMES:
Decrease in relapse rate | 3 months after dislocation
  Evidence of a significant decrease in the relapse rate when the arm is immobilized in an external rotation position
Decrease in relapse rate | 12 months after dislocation
  Evidence of a significant decrease in the relapse rate when the arm is immobilized in an external rotation position
Decrease in relapse rate | 24 months after dislocation
  Evidence of a significant decrease in the relapse rate when the arm is immobilized in an external rotation position

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pelet, MD, PhD, Principal Investigator — Hôpital Enfant-Jésus
Locations (1):
- CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada